CLINICAL TRIAL: NCT02526147
Title: WFP Cash, Food, and Voucher Study in Ecuador
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: World Food Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 6119-001
Record Dates: First submitted 2015-08-12; First posted 2015-08-18 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Food Security
MeSH Terms: interventions — CASP8 and FADD-Like Apoptosis Regulating Protein; Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): Receives no intervention
- Cash (Experimental): Household receives cash transfer monthly for 6 months
  Interventions: Other: Cash
- Voucher (Experimental): Household receives food voucher to use at local supermarket monthly for 6 months
  Interventions: Other: Voucher
- Food (Experimental): Household receives food transfer composed of rice, lentils, canned sardines, and vegetable oil, monthly for 6 months
  Interventions: Other: Food

INTERVENTIONS:
Other: Cash
  Arms: Cash
Other: Voucher
  Arms: Voucher
Other: Food
  Arms: Food

SUMMARY:
This evaluation is part of a five country project to evaluate the benefits and costs of the use of two alternatives to food transfers: vouchers and cash (hereafter referred to as "alternative modalities"). The project will generate information on how outcomes such as household food expenditure and dietary diversity, relevant to both beneficiaries and WFP, change following the introduction of these alternative modalities; how benefits and costs of these are, relative to food transfers, distributed across and within households; and what are the critical operational issues that need to be addressed for these alternatives to be successfully implemented. More specifically, the project will answer seven questions:

1. Do households benefit from receipt of the alternative modalities?
2. Are these benefits greater, or less, when transfers are made using alternative modalities compared to food transfers. How does this vary across outcomes (such as nutrition, livelihoods, gender dynamics and intra-household resource allocation) that are of especial interest to WFP?
3. How does the distribution of benefits differ across households when transfers are made using alternative modalities compared to food transfers?
4. How does the distribution of benefits differ within households when transfers are made using alternative modalities compared to food transfers? Do certain household members (women, young children) benefit more from one type of modality? How do these modalities affect decision-making processes within the household?
5. Why are these differences observed? How do the reasons for these differences affect the study's ability to generalize from these evaluations?
6. Does the delivery of alternative modalities cost less than food transfers? What accounts for these cost differences? Are some costs (such as transport) really lower or are they transferred to beneficiaries? Within the household, who bears these additional costs?
7. What is the benefit: cost ratios associated with these different modalities from the perspective of WFP? Is there a conflict between the modality "preferred" by WFP and the modality "preferred" by beneficiaries?

These objectives will be accomplished through household survey data collection among a panel of households before and after transfer of alternative modalities. In addition, select countries will involve the collection of anthropometric, biomarker and cognitive testing.

DETAILED DESCRIPTION:
In Ecuador, the intervention consists of food, food vouchers or cash transfers to Colombian refugees and poor Ecuadorian households in four urban and peri-urban areas of Carchi and Sucumbios in northern Ecuador. The transfer is given monthly for 6 months. The program is conditional on attendance at nutrition and community trainings occurring once a month. In most cases the transfer recipient is the female head of household or spouse, however in some cases men may also receive the transfer.

The study is a 2 stage randomized control trial where, first, 80 neighborhoods were randomized to either treatment or control group; second, treatment clusters (geographical units within neighborhoods) were randomized to either: cash, food voucher or food assistance. Approximately 20 - 28 participants from each of the 145 clusters were randomly selected for interviews. In addition to the household socio-economic survey, hemoglobin measures were taken from children between 6 months and 5 years of age and adolescent girls from age 10 to 16 years in each household. The baseline survey occurred in April 2011 and the endline in November 2011.

Interviews were conducted with female heads of households or spouses where possible, or with adult male head of households. In addition, hemoglobin was collected for all children ages 6 months to 5 years and for adolescent girls residing in surveyed households.

ELIGIBILITY:
Inclusion Criteria:

* Households in pre-selected neighborhoods in Carchi and Sucumbios with high poverty status according to the proxy means test.
* For hemoglobin measurements, children residing in these households that are 6 months-5 years old, and adolescent girls 10-16 years old

Exclusion Criteria:

* Households that receive the Bono de Desarrollo Humano
* Children ages 6 months - 5 years who are severely sick

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2580 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Food security as measured by the value of food consumption through a household questionnaire | 6 months
  Value of food consumption is a monetary value greater than zero of food consumed in the household in the last week.
Dietary diversity as measured by dietary diversity index and food consumption score through a household questionnaire | 6 months
  Dietary diversity index is the number of food items consumed in the household in the last week. Household questionnaire asks about 41 food items, and thus the index ranges from 0-41.
  Food consumption score uses same information from food items consumed in the last week, groups them into 8 food groups (staples, pulses, vegetables, fruit, meat/fish, milk/dairies, sugar/honey, oils/fats), sums the number of days these eight different food groups were consumed, and then weights the different groups according to their nutritional value. The score ranges from 0-112.

SECONDARY OUTCOMES:
Mean hemoglobin level as measured by a portable hemoglobinometer (Hemocue AB, Sweden) | 6 months
  Hemoglobin concentration of whole blood will be determined using a portable hemoglobinometer (Hemocue AB, Sweden); a single drop of whole capillary blood from the tip of the middle or index finger will be transferred to the microcuvette using a glass pipette and results will be recorded to the nearest 1 g/L.
Prevalence of intimate partner violence as measured by WHO Violence Against Woman Instrument | 6 months
  Measures the percent of women who have experienced physical violence, controlling behaviors, or emotional violence.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa L Hidrobo, PhD, Principal Investigator — IFPRI

REFERENCES:
- [Derived] Buller AM, Hidrobo M, Peterman A, Heise L. The way to a man's heart is through his stomach?: a mixed methods study on causal mechanisms through which cash and in-kind food transfers decreased intimate partner violence. BMC Public Health. 2016 Jun 8;16:488. doi: 10.1186/s12889-016-3129-3. PMID 27278935